CLINICAL TRIAL: NCT02223286
Title: Understanding Clinician Utilization of Corus CAD (Age/Sex/Gene Expression Score - ASGES) in Clinical Decision Making
Acronym: UCU-CARD
Status: Completed | Type: Observational
Sponsor: CardioDx (Industry)
Responsible Party: Sponsor
Other Study IDs: CDX_000016; UCU-CARD (Other: CardioDx)
Record Dates: First submitted 2014-08-19; First posted 2014-08-22 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Coronary Artery Disease; Angina Pectoris; Chest Pain; Cardiovascular Diseases; Coronary Heart Disease; CAD; CVD; CHD
Keywords: Corus CAD; ASGES; Age/Sex/Gene Expression Score; Gene Expression; GES; CAD; CVD; CHD; Precision Medicine; Clinical Utility; Coronary Artery Disease; Angina Pectoris; Chest Pain; Cardiovascular Disease; Coronary Heart Disease; UCU-CARD
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Chest Pain; Cardiovascular Diseases; Coronary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ASGES (Treatment Group): Patients who received a Corus CAD or Age/Sex/Gene Expression Score (ASGES) to aid in the diagnosis of obstructive CAD
  Interventions: Diagnostic Test: Corus CAD
- Non-ASGES (Control Group): Patients who underwent usual care testing and did not receive a Corus CAD or Age/SEX/Gene Expression Score (ASGES) to aid in the diagnosis of obstructive CAD

INTERVENTIONS:
Diagnostic Test: Corus CAD — Age/Sex/Gene Expression Score
  Groups: ASGES (Treatment Group)

SUMMARY:
The purpose of this study is to understand the use of Corus CAD also known as Age/Sex/Gene Expression score (ASGES) in the clinical decision making process of patients who underwent the evaluation of chest pain or anginal equivalent symptoms. Specifically, to better understand whether the use of the assay in clinical decision making resulted in changes in noninvasive diagnostic test ordering or diagnostic yield of additional tests ordered and/or invasive angiography.

DETAILED DESCRIPTION:
The UCU-CARD (Understanding Clinician Utility-Cardiology) study is a retrospective, matched-cohort evaluation of diagnostic testing in a community-based cardiology practice setting that used a personalized age, sex, and gene expression test during early work-up of patients with symptoms suggestive of obstructive CAD (http://www.clinicaltrials.gov, NCT02223286). The study measured the rates of advanced cardiac diagnostic testing after initial work-up, including stress testing with imaging, CTA, or ICA. Rates of advanced diagnostic testing for patients who received the age, sex, and gene expression test (ASGES) were compared with testing rates for matched historical controls (usual care). The study hypothesis was that incorporating the age, sex, and gene expression testing early in the diagnostic work-up pathway would permit the identification of patients for whom advanced diagnostic testing was not required, thereby avoiding unnecessary testing and enabling cardiologists to focus their diagnostic resources more efficiently.

This single-center study was conducted at the North Phoenix Heart Center (Phoenix, AZ), a community-based group cardiology practice that receives patients on referral from primary care physicians and other specialists in the surrounding area. The practice incorporated age, sex, and gene expression testing into its diagnostic protocol beginning in June 2011. Data collection was completed in December 2013. Institutional Review Board (IRB) approval of the study protocol was granted by Quorum Review. Informed consent waivers were granted as data collection was retrospective and all data were de-identified.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms suggestive of CAD, according to the opinion of the site clinician
2. Age >= 21 years

Exclusion Criteria:

1. History of myocardial infarction (MI)
2. History of high risk unstable angina, systemic infections or systemic inflammatory conditions
3. Current MI or acute coronary syndrome
4. Current New York Heart Association (NYHA) class III or IV congestive heart failure symptoms
5. Known/documented CAD
6. History/current Diabetes Mellitus
7. Taking steroids, immunosuppressive agents, or chemotherapeutic agents, at time of chest pain presentation

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population of interest and the main inclusion criterion for inclusion is the occurrence of chest pain (or anginal equivalent) in a patient without known significant CAD or a history of prior myocardial infarction, and the utilization of Corus CAD (Age/Sex/Gene Expression score - ASGES).
  Additionally, subjects with similar chest pain (or angina equivalent) whom did not undergo Corus CAD (ASGES) will be included as a control group, to understand the diagnostic evaluation and management of patients prior to Corus CAD (ASGES) use.
Sampling Method: Non-Probability Sample
Enrollment: 552 (Actual)
Dates: Start 2013-03; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The primary measure of this study is the number of advanced diagnostic tests in ASGES (treatment group) patients compared to the number of advanced diagnostic tests in non-ASGES (control group) patients. | up to 24 months
  The primary study endpoint was the percentage of patients for whom advanced diagnostic testing was ordered-stress testing with imaging, computed tomography angiography, or invasive coronary angiography.

CONTACTS AND LOCATIONS:
Overall Officials: David Hoffman, DO, Principal Investigator — Northeast Ohio Medical University; Lawrence Kline, DP, Principal Investigator — John C. Lincoln Heart Institute; Jaime Burkle, MD, Principal Investigator — Piedmont Heart Institute
Locations (3):
- United States (3):
  - John C. Lincoln Heart Institute, Phoenix, Arizona
  - Piedmont Heart Institute, Blue Ridge, Georgia
  - Heart Associates, Youngstown, Ohio